CLINICAL TRIAL: NCT05010174
Title: Extension Study to Assess the Long-Term Safety in Recipients Who Previously Received Medeor's Cellular Immunotherapy Products
Brief Title: Long-term Safety Follow-up in Recipients Who Previously Received Medeor's Cellular Immunotherapy Products
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Medeor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDR-105-SAE
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Immune Tolerance
Keywords: Long-term follow-up

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational, long-term safety follow-up of patients who have received MDR product: Only patients who have received treatment with MDR product will be eligible for this study.
  Interventions: Drug: MDR product

INTERVENTIONS:
Drug: MDR product — Observation of patients previously receiving MDR product(s)

SUMMARY:
At the completion of primary follow-up of various Medeor Transplant studies (called parent studies), subjects receiving Medeor's cellular immunotherapy products will be followed annually for up to an additional 84 months (7 years), in order to evaluate for long-term safety.

DETAILED DESCRIPTION:
Study MDR-105-SAE is intended to be the long-term safety monitoring extension of Medeor's cellular immunotherapy, kidney transplant clinical studies. This Master Protocol has been created in order to establish a single database for all long-term safety data for those subjects that have received Medeor's cellular products. This Master Protocol will provide up to 84 months (7 years) of additional follow-up.

Long-term safety of subjects treated with Medeor's cellular immunotherapy has not been assessed. This study will collect the data into a centralized database allowing for continuous monitoring of any important safety signals.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to fully comply with all study procedures and restrictions.
2. Able to understand and provide written, signed, and dated informed consent to participate in the study in accordance with ICH GCP Guideline and all applicable local regulations.
3. Have previously completed a Medeor study and received a Medeor cellular immunotherapy product

Exclusion Criteria:

1. Has any condition or circumstance, which in the opinion of the Investigator would significantly interfere with the subject's protocol compliance or put the subject at increased risk.
2. Unable or unwilling to provide written, signed, and dated informed consent to participate in the study.
3. Has undergone a second organ transplant with an organ derived from an individual other than the donor of the transplant kidney received during a Medeor study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients who received Medeor's cellular immunotherapy in previous Medeor studies
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints | Through study completion, up to 7 years
  Incidence of serious adverse events (SAEs), adverse events (AEs) leading to study withdrawal, and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Lenuta Micsa, MD, Study Director — Medeor Therapeutics
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided